CLINICAL TRIAL: NCT00002763
Title: POST-OPERATIVE ADJUVANT INTERFERON-ALFA-2B (INTRON-A) TREATMENT AFTER RESECTION OF THICK PRIMARY MELANOMA AND/OR REGIONAL LYMPHNODE METASTASES 'INTERMEDIATE-HIGH DOSE' VS INTERMEDIATE-LOW DOSE' IFN-ALFA VS OBSERVATION: A 3-ARM MULTICENTER RANDOMIZED PHASE III TRIAL
Brief Title: High-Dose or Low-Dose Interferon Alfa Compared With No Further Therapy Following Surgery in Treating Patients With Stage III Melanoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064718; EORTC-18952
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Interferon-alpha

INTERVENTIONS:
Biological: recombinant interferon alfa

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells. It is not known whether giving high-dose or low-dose interferon alfa is more effective than no further therapy in treating patients with stage III melanoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of high- or low-dose interferon alfa with that of no further therapy following surgery in treating patients who have stage III melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the time to distant metastasis, death due to melanoma, and overall survival in patients with high-risk stage III melanoma treated with 10 MU of interferon alfa (IFN-A) for 4 weeks followed by 1 year of IFN-A at 10 MU three times per week vs. 2 years of IFN-A at 5 MU three times per week vs. observation alone. II. Assess the toxicity associated with IFN-A. III. Compare the quality of life, costs, and compliance associated with each treatment regimen.

OUTLINE: Randomized study. Following definitive surgical resection, patients are randomly assigned in a 2:2:1 ratio to Arms A, B, and C, respectively. Arm A: Biological Response Modifier Therapy. Interferon alfa-2b (Schering), IFN-A, NSC-377523. Higher dose. Arm B: Biological Response Modifier Therapy. IFN-A. Lower dose. Arm C: Control. Observation.

PROJECTED ACCRUAL: A total of 1,000 patients will be entered over approximately 4 years in this multicenter study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Cutaneous melanoma in one of the following categories: T4, N0, M0 Deep primary tumor with Breslow depth greater than 4.0 cm Tx, N1, M0 Primary tumor with regional lymph node metastases found at lymphadenectomy but clinically undetectable Tx, N2, M0 Clinically apparent regional lymph node metastases (synchronous or metachronous) confirmed by lymphadenectomy Definitive surgical resection and lymphadenectomy with pathologically confirmed adequate surgical margins required Minimum 2 cm margin for primary lesions with Breslow depth greater than 2 mm Distal interphalangeal amputation required for subungual melanomas No primary melanoma originating apart from the skin No multiple in transit metastases in an extremity No lymph node involvement outside the operative area resected by radical neck, axillary lymph node, or ilioinguinal dissection

PATIENT CHARACTERISTICS: Age: 16 to 75 Performance status: ECOG 0 or 1 Hematopoietic: WBC at least 4,000 Platelets at least 125,000 Hemoglobin at least 9.8 g/dL (6.1 mmol/L) Hepatic: Bilirubin no greater than 2 times normal AST no greater than 2 times normal Renal: Creatinine no greater than 1.6 mg/dL (140 micromoles/L) Cardiovascular: No ventricular or supraventricular arrhythmia requiring treatment No congestive heart failure (NYHA class 3/4 status) Other: No uncontrolled infection No requirement for ongoing steroids, NSAIDs, or other immunomodulators No organic brain syndrome or significant impairment of basal cognitive function No psychiatric disorder that would preclude study participation or would be exacerbated by study therapy (e.g., depression) No second malignancy except: In situ cervical cancer Nonmelanomatous skin cancer No pregnant or nursing women

PRIOR CONCURRENT THERAPY: No prior treatment on this protocol for patients with recurrent melanoma at regional lymph nodes No preoperative infusion or perfusion therapy Biologic therapy: No prior adjuvant immunotherapy Chemotherapy: No prior adjuvant systemic chemotherapy No prior anthracyclines Endocrine therapy: Not specified Radiotherapy: No prior adjuvant radiotherapy Surgery: See Disease Characteristics

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 1996-04

CONTACTS AND LOCATIONS:
Overall Officials: Alexander M. M. Eggermont, MD, PhD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center
Locations (86):
- Austria (2):
  - Krankenhaus der Elisabethinen, Linz
  - Landeskrankenanstalten - Salzburg, Salzburg
- Belgium (7):
  - Hopital Universitaire Erasme, Brussels
  - Institut Jules Bordet, Brussels (Bruxelles)
  - Cliniques Universitaires Saint-Luc, Brussels (Bruxelles)
  - Centre Hospitalier Notre Dame - Reine Fabiola, Charleroi
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent (Gent)
  - U.Z. Gasthuisberg, Leuven
- Bulgaria (2):
  - Alexander's University Hospital, Sofia
  - National Centre of Oncology, Sofia
- University Hospital Sestre Milosrdnice, Zagreb, Croatia
- Estonian Cancer Center, Tallinn, Estonia
- Finland (2):
  - Tampere University Hospital, Tampere
  - Turku University Central Hospital, Turku
- France (19):
  - CHU de Bordeaux - Hopital Pellegrin, Bordeaux
  - Institut Bergonie, Bordeaux
  - CHU Ambroise Pare, Boulogne-Billancourt
  - CHRU de Caen, Caen
  - Centre Leon Berard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Hopital L'Archet - 2, Nice
  - Hopital Bichat-Claude Bernard, Paris
  - Hopital Saint-Louis, Paris
  - Hopital Cochin, Paris
  - Hopital Haut Leveque, Pessac
  - Centre Eugene Marquis, Rennes
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Hospitalier Regional et Universitaire de Saint-Etienne, Saint-Priest-en-Jarez
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Centre Hospitalier Regional Metz Thionville, Thionville
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Institut Gustave Roussy, Villejuif
- Germany (14):
  - Universitaetsklinikum Benjamin Franklin, Berlin
  - Robert Roessle Klinik, Berlin
  - Universitaets-Augenklinik - Erlangen, Erlangen
  - Georg August Universitaet, Göttingen
  - Universitats-Krankenhaus Eppendorf, Hamburg
  - Haematologisch-Onkologische Praxis Altona, Hamburg
  - Department of Dematology, Hannover Medical School, Hanover
  - Universitaets-Hautklinik Heidelberg, Heidelberg
  - Universitatsklinik, Saarland, Homburg/Saar
  - III Medizinische Klinik Mannheim, Mannheim
  - Klinikum der Universitat Regensburg, Regensburg
  - Universitatshautklinik Eberhard - Karlsuniversitat Tubingen, Tübingen
  - Department of Dermatology, Ulm
  - Universitaet Wuerzburg/Hautkrankheiten, Würzburg
- Israel (2):
  - Wolfson Medical Center, Holon
  - Tel-Aviv Medical Center-Ichilov Hospital, Tel Aviv
- Istituto Europeo Di Oncologia, Milan, Italy
- Netherlands (7):
  - Academisch Ziekenhuis der Vrije Universiteit, Amsterdam
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - University Medical Center Nijmegen, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
  - Academisch Ziekenhuis Utrecht, Utrecht
- Poland (3):
  - Medical University of Gdansk, Gdansk
  - Maria Sklodowska-Curie M.C.C.I.O. Krakow, Krakow (Cracow)
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw
- Portugal (2):
  - Instituto Portugues de Oncologia de Francisco Gentil, Lisbon
  - Instituto Portugues de Oncologia do Porto, Porto
- Russian Academy of Medical Sciences Cancer Research Center, Moscow, Russia
- Institute of Oncology and Radiology of Serbia, Belgrade, Serbia
- National Cancer Institute - Bratislava, Bratislava, Slovakia
- Spain (2):
  - Hospital Clinic y Provincial de Barcelona, Barcelona
  - Hospital Clinico Universitario, Zaragoza
- Huddinge Hospital, Huddinge, Sweden
- Switzerland (6):
  - Ospedale San Giovanni, Bellinzona
  - Inselspital, Bern, Bern
  - Ratisches Kantons und Regionalspital, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital - Saint Gallen, Sankt Gallen
  - Universitaetsspital, Zurich
- Turkey (Türkiye) (5):
  - Cukurova University School of Medicine, Adana
  - Vakif Gureba Training Hospital, Istanbul
  - Istanbul University-Institute of Oncology, Istanbul
  - Cerrahpasa Medical School, Istanbul
  - Ege University Medical School, Izmir
- United Kingdom (6):
  - Bristol Oncology Centre, Bristol, England
  - Addenbrooke's NHS Trust, Cambridge, England
  - St. James's Hospital, Leeds, England
  - Royal Marsden NHS Trust, London, England
  - Derriford Hospital, Plymouth, England
  - Beatson Oncology Centre, Glasgow, Scotland

REFERENCES:
- [Background] Eggermont AM, Suciu S, Testori A, Kruit WH, Marsden J, Punt CJ, Santinami M, Sales F, Schadendorf D, Patel P, Dummer R, Robert C, Keilholz U, Yver A, Spatz A. Ulceration and stage are predictive of interferon efficacy in melanoma: results of the phase III adjuvant trials EORTC 18952 and EORTC 18991. Eur J Cancer. 2012 Jan;48(2):218-25. doi: 10.1016/j.ejca.2011.09.028. Epub 2011 Nov 5. PMID 22056637
- [Background] Bouwhuis MG, Suciu S, Collette S, Aamdal S, Kruit WH, Bastholt L, Stierner U, Sales F, Patel P, Punt CJ, Hernberg M, Spatz A, ten Hagen TL, Hansson J, Eggermont AM; EORTC Melanoma Group and the Nordic Melanoma Group. Autoimmune antibodies and recurrence-free interval in melanoma patients treated with adjuvant interferon. J Natl Cancer Inst. 2009 Jun 16;101(12):869-77. doi: 10.1093/jnci/djp132. Epub 2009 Jun 9. PMID 19509353
- [Background] Eggermont AM, Punt CJ. Does adjuvant systemic therapy with interferon-alpha for stage II-III melanoma prolong survival? Am J Clin Dermatol. 2003;4(8):531-6. doi: 10.2165/00128071-200304080-00002. PMID 12862495
- [Result] Bouwhuis MG, Collette S, Suciu S, de Groot ER, Kruit WH, Ten Hagen TL, Aarden LA, Eggermont AM, Swaak AJ; EORTC Melanoma Group. Changes of ferritin and CRP levels in melanoma patients treated with adjuvant interferon-alpha (EORTC 18952) and prognostic value on treatment outcome. Melanoma Res. 2011 Aug;21(4):344-51. doi: 10.1097/CMR.0b013e328346c17f. PMID 21546857
- [Result] Bouwhuis MG, Suciu S, Kruit W, Sales F, Stoitchkov K, Patel P, Cocquyt V, Thomas J, Lienard D, Eggermont AM, Ghanem G; European Organisation for Research and Treatment of Cancer Melanoma Group. Prognostic value of serial blood S100B determinations in stage IIB-III melanoma patients: a corollary study to EORTC trial 18952. Eur J Cancer. 2011 Feb;47(3):361-8. doi: 10.1016/j.ejca.2010.10.005. Epub 2010 Nov 17. PMID 21087856
- [Result] Bouwhuis M, Suciu S, Kruit W, et al.: Prognostic value of autoantibodies (auto-AB) in melanoma patients (pts) in the EORTC 18952 trial of adjuvant interferon (IFN) compared to observation (obs). [Abstract] J Clin Oncol 25 (Suppl 18): A-8507, 473s, 2007.
- [Result] Suciu S, Ghanem G, Kruit W, et al.: Serum S-100B protein is a strong independent prognostic marker for distant-metastasis free survival (DMFS) in stage III melanoma patients: an evaluation of the EORTC randomized trial 18952 comparing IFNα versus observation. [Abstract] J Clin Oncol 25 (Suppl 18): A-8518, 476s, 2007.
- [Result] Eggermont AM, Suciu S, MacKie R, Ruka W, Testori A, Kruit W, Punt CJ, Delauney M, Sales F, Groenewegen G, Ruiter DJ, Jagiello I, Stoitchkov K, Keilholz U, Lienard D; EORTC Melanoma Group. Post-surgery adjuvant therapy with intermediate doses of interferon alfa 2b versus observation in patients with stage IIb/III melanoma (EORTC 18952): randomised controlled trial. Lancet. 2005 Oct 1;366(9492):1189-96. doi: 10.1016/S0140-6736(05)67482-X. PMID 16198768